CLINICAL TRIAL: NCT02337790
Title: Necklace-Shaped Sensor for Non-Invasive Monitoring of Fluids, Heart Rate, Heart Rate Variability, and Respiration Rate in Patients With a Pacemaker, Implanted Cardioverter-Defibrillator, or Ventricular Assist Device
Brief Title: Necklace-Shaped Sensor for Non-Invasive Remote Monitoring of Vitals
Status: Completed | Type: Observational
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: PERM-IRB-001-ICC
Record Dates: First submitted 2015-01-09; First posted 2015-01-14 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Heart Failure; Hypertension
Keywords: Hypertension; Heart Failure; Fluids
MeSH Terms: conditions — Heart Failure; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort 1: Subjects will have a pacemaker, implanted cardioverter-defibrillator, or ventricular assist device.

SUMMARY:
This study is designed to validate the use of the CoVa Monitoring System in subjects with implanted devices.

DETAILED DESCRIPTION:
The study had the following objectives:

1. Verify that the CoVa Monitoring System does not interfere with implanted devices.
2. Verify that implanted devices do not interfere with the functions of the CoVa Monitoring System.
3. Verify that the CoVa Monitoring System fits on a wide variety of body types.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between 21 (twenty-one) and 95 (ninety-five) years of age at screening.
* Subject has a pacemaker, implanted cardioverter-defibrillator, or ventricular assist device.
* Subject and/or legally authorized person/representative is willing to undergo the Informed Consent process prior to enrollment in the study.
* Subject is a candidate for this study based on the PI's opinion and knowledge of the subject's condition.

Exclusion Criteria:

* Subject is participating in another clinical study that may affect the results of either study.
* Subject is unable or not willing to wear electrode patches as required.
* Subject has skin sensitivity to adhesive or hydrogel materials used in electrode patches.
* Subject is considered by the PI to be medically unsuitable for study participation.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be from the Imperial Cardiac Clinic
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2015-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Interference between implanted devices and CoVa Monitoring System | One time for up to 15 minutes during a clinic visit for device interrogation

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Banet, PhD, Principal Investigator — Baxter Healthcare Corporation
Locations (1):
- Imperial Cardiac Center, Imperial, California, United States